CLINICAL TRIAL: NCT05972746
Title: Telemonitoring Program With Electronic Alerts to Improve Outcomes in the Vulnerable Phase After Hospitalization for Heart Failure: A Pragmatic Clinical Trial TREAT - Vulnerable HF
Brief Title: Telemonitoring Program in the Vulnerable Phase After Hospitalization for Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Cardiovascular de Buenos Aires (Other)
Responsible Party: Principal Investigator, Lucrecia Maria Burgos, Unit coordinator, Instituto Cardiovascular de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0
Record Dates: First submitted 2023-04-14; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Acute Heart Failure
Keywords: telemonitoring; Heart Failure; Vulnerable phase
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring program with electronic alerts + Standard of care (Experimental)
  Interventions: Device: Telemonitoring with electronic alerts; Other: Standard of care
- Standard of care (Placebo Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Telemonitoring with electronic alerts — Patients assigned to this group will receive standard care plus a telemonitoring program.
  Arms: Telemonitoring program with electronic alerts + Standard of care
Other: Standard of care — Standard of care

SUMMARY:
This pragmatic clinical trial aims to evaluate the impact of a telemonitoring program with an electronic alert system compared to standard treatment on the perception of self-care in patients after hospitalization for decompensated HF at 3 months post-discharge. And secondarily to evaluate its impact on clinical events, NT-proBNP and efficacy and safety to facilitate the use and titration of the recommended drugs in patients with reduced ejection fraction at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized for acute heart failure (regardless of the level of left ventricular ejection fraction) within 24 hours of discharge, or with a history of hospitalization for acute HF within 10 days prior to randomization.
* Own a smartphone (Smartphone) with internet Ability to speak and read Spanish.
* Residence in the metropolitan area of Buenos Aires

Exclusion Criteria:

* Pregnancy
* Alcohol or drug abuse
* Kidney failure in hemodialysis,
* Inability to use the app (Ex: cognitive impairment, lack of social support, lack of ability to communicate)
* Active cancer
* Life expectancy less than 1 year
* Candidates for care home or institutional end of life
* Severe psychiatric illness
* Planned cardiac surgery
* Patient unable or unwilling to give informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-10-07 (Estimated); Study Completion 2023-11-07 (Estimated)

PRIMARY OUTCOMES:
Self-care behavior | 90 days
  The EHFScBS scale will be used. It consists of a self-administered questionnaire with 12 items addressing various aspects of patient self-care. Each item is scored from 1 (completely agree/always) to 5 (completely disagree/never). The overall score can range from 12 (best self-care) to 60 (worst self-care)

SECONDARY OUTCOMES:
NT pro BNP | 90 days
Medication adherence | 90 days
Quality of life | 90 days
  The specific Quality of Life (QoL) related to heart failure will be assessed using the Minnesota Living with Heart Failure Questionnaire (MLHFQ), which consists of 21 items. Participants rate their perceptions of how heart failure and its treatment affect their daily life on a 6-point Likert scale ranging from 0 (no impairment) to 5 (very impaired). Therefore, lower scores indicate better specific QoL related to heart failure, and a change of 5 points is considered the minimum clinically significant change [30]. The MLHFQ yields a total QoL score and separate scores for the physical and emotional well-being sub-scales.
First readmission for heart failure | 90 days
Total number of readmissions for heart failure | 90 days
Time to achieve the use of Guideline-Directed Medical Therapy | 90 days
Proportion of patients with heart failure and reduced ejection fraction who have an increase in the number of Guideline-Directed Medical Therapy | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Cardiovascular de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided